CLINICAL TRIAL: NCT03146039
Title: Non-Invasive Cervical Cancer Radiotherapy: Phase II Clinical Trial of Stereotactic Body Radiotherapy Boost for Stage IB-IVB Cervical Cancer
Brief Title: Non-Invasive Cervical Cancer Radiotherapy for Stage IB-IVB
Acronym: NICER
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Patient enrollment goal will not be met
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Loren Mell, MD, Associate Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSD 161328
Record Dates: First submitted 2017-04-25; First posted 2017-05-09 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Cervical Cancer; Cervical Cancer Stage; Cervical Cancer Stage IB2; Cervical Cancer Stage IB1; Cervical Cancer Stage I; Cervical Cancer Stage IB; Cervical Cancer Stage II; Cervical Cancer Stage IIa; Cervical Cancer, Stage IIB; Cervical Cancer, Stage III; Cervical Cancer Stage IIIB; Cervical Cancer Stage IIIA; Cervical Cancer Stage Iv; Cervical Cancer Stage IVA; Cervical Cancer Stage IVB
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Radiation Therapy (Other): The patient will receive Whole Pelvis Radiation Therapy 40 - 50.4 Gy in 1.8 - 2.0 Gy daily fractions over 4.5 - 5.5 weeks followed by Stereotactic Body Radiotherapy 5.5 - 8.0 Gy per fraction x 5 fractions using arc therapy.
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Whole pelvis radiation therapy will be delivered according to institutional standard of care.
  SBRT is delivered with 5 fractions of 5.5-8 Gy prescribed to the high-risk CTV, with dose constraints identical to those for high dose rate, volume-directed brachytherapy. The patient will undergo arc therapy with a minimum of two arcs. On-line kV CBCT will be used to verify the isocenter prior to each arc delivery. Patients will be resimulated for SBRT boost planning.

SUMMARY:
The purpose of this study is to find out whether patients with cervical cancer treated with about a new radiation technique called "stereotactic body radiotherapy (SBRT) have less stress and anxiety compared to standard brachytherapy radiation. With standard brachytherapy radiation, metal hardware is placed through the vagina and into the uterus, which can cause pain and discomfort. SBRT is a new radiation technique that is non-invasive and does not require the insertion of any metal hardware.

DETAILED DESCRIPTION:
This is a Phase II, single-center, single-arm, study of Stereotactic Body Radiotherapy boost for stage IB-IVB cervical cancer.

The primary objective of the study is to test the hypothesis that stereotactic body radiation therapy (SBRT) leads to an improvement in treatment-related symptoms of post traumatic stress compared to brachytherapy (historical control) according to the Impact of Event Scale-Revision (IES-R).

Study participants will be recruited within the UCSD Health System. For those patients under the clinical management of the recruiting investigator, the investigator will review the patient's medical records and determine if they would be a candidate for the study. The investigator will approach the subject and offer participation in the trial. If the patient chooses to participate, they will undergo pretreatment evaluations to determine if they are a good candidate to participate further in the study. Depending on when the patient last had these tests and procedures performed, some of them may not need to be repeated.

Upon confirmation of all eligibility criteria, the subject will be enrolled. Each enrolled subject will receive radiation therapy consisting of 30 to 35 treatments. The patient will first undergo Whole Pelvis Radiation Therapy 40 - 50.4 Gy in 1.8 - 2.0 Gy daily fractions over 4.5 - 5.5 weeks, followed by Stereotactic Body Radiotherapy 5.5 - 8.0 Gy per fraction x 5 fractions using arc therapy. Concurrent chemotherapy may be given with radiation therapy according to the discretion of the treating oncology team. No chemotherapy will be given during the SBRT phase of treatment. During radiation therapy, the patient will have a weekly physical exam, vital signs collected, evaluation for pain, and review any side effects.

Subjects will undergo a post treatment follow-up period after completion of their radiation therapy. During this follow-up period, subjects will return for a medical and history review with a complete physical examination, review of any side effects, evaluation for outcomes and toxicity, and evaluations for stress, anxiety, and pain.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven, invasive carcinoma of the cervix.
* Candidate for pelvic, pelvic-inguinal, or extended field radiotherapy with or without concurrent chemotherapy. Patients undergoing preoperative or adjuvant chemotherapy are excluded.
* History/physical examination within 60 days prior to registration to document cervical tumor size and stage
* CT, MRI, or PET/CT imaging of the chest, abdomen, and pelvic regions within 60 days prior to registration (for stage I patients, PA and lateral chest x-ray is sufficient for chest imaging)
* Age ≥ 18
* Negative serum pregnancy test for women of child-bearing potential
* Women of childbearing potential must agree to practice effective birth control throughout their participation in the treatment phase of the study.
* Patients must sign informed consent prior to study entry.

Exclusion Criteria:

* Prior radiotherapy to the pelvis or abdomen that would result in overlap of radiation therapy fields.
* Prior hysterectomy.
* Women who are pregnant or lactating are ineligible due to teratogenic effects on developing fetuses. Women who are of child-bearing potential need to practice effective methods of contraception including oral contraceptives, intrauterine device, diaphragm with spermicides, and/or abstinence.
* Patients undergoing preoperative or adjuvant chemotherapy
* History of pre-existing PTSD.
* History of major psychiatric disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Number of Treatment-Related Symptoms of Post Traumatic Stress | 2 years
  To quantify treatment-related symptoms of post traumatic stress to determine if stereotactic body radiation therapy (SBRT) leads to an improvement in treatment-related symptoms of post traumatic stress compared to brachytherapy (historical control) according to the Impact of Event Scale-Revision (IES-R).

SECONDARY OUTCOMES:
Number of Patients with Adverse Events Following SBRT as a Measure of Safety | 2 years
  To quantify rates of acute hematologic, gastrointestinal, and genitourinary toxicity following SBRT.
Ranking Quality of Life of Patients | 2 years
  To measure health-related quality of life based on the cancer-specific EORTC-QLQ-C30 questionnaire (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30).
Ranking Quality of Life of Patients | 2 years
  To measure health-related quality of life based on the cervical cancer module (CX24).
Number of Intrafraction Cervical Motion | 2 years
  To quantify intrafraction cervical motion using cone beam computed tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Loren Mell, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Moores UC San Diego Cancer Center, La Jolla, California, United States